CLINICAL TRIAL: NCT06887309
Title: Cerebral Reorganizations Induced by Spinal Cord Injury Spinal Cord Injury: Multimodal Assessments of Sensory-motor and Cognitive-behavioral Functions. SUPRASPINAL
Brief Title: Spinal Cord Injury: Impact on Sensory, Motor, Behavioral and Cognitive Functions
Acronym: SUPRASPINAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL23_0434; 2024-A00206-41 (Other: ANSM)
Record Dates: First submitted 2025-02-07; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; fMRI; DTI; MRI; diffusion tensor imaging
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients spinal cord injury with incomplete sensorimotor deficits ( ASIA B, C, D) and with complete (Experimental): Experimental: Patients spinal cord injury with incomplete sensorimotor deficits (ASIA B, C, D) and with complete sensorimotor deficits (ASIA A)
  Interventions: Diagnostic Test: MRI; Behavioral: Neuropsychological tests
- Healthy control group (Active Comparator): MRI : anatomical (3DT1, 3D-FLAIR), functional (task-based and resting-state) and tractographic (multiband diffusion imaging). MRI will be done once for the healthy volunteer control group.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI : anatomical (3DT1, 3D-FLAIR), functional (task-based and resting-state) and tractographic (multiband diffusion imaging) at three time points: one week, three months and twelve months after the spinal cord injury (SCI)
Behavioral: Neuropsychological tests — The following tests will be performed: the Montreal Cognitive Assessment (MOCA), the Montgomery-Åsberg depression rating scale (MADRS), the Medical Outcome Study Short Form 36 (SF-36)
  Arms: Patients spinal cord injury with incomplete sensorimotor deficits ( ASIA B, C, D) and with complete

SUMMARY:
Spinal cord injury (SCI) causes a variety of sensory-motor deficits and neuropsychological consequences. Magnetic resonance imaging (MRI) reveals a reduction in the volume of the somato-sensory and motor cortices, as well as atrophy in the white matter bundles. In addition, disturbances in cerebral activity are observed in several areas, notably the motor cortex and the prefrontal cortex. The aim of this study is to understand the evolution of brain function after SCI in comparison with a control group of healthy volunteers.

We distinguish between patients with incomplete sensorimotor deficits (ASIA B,C,D) and complete sensorimotor deficits (ASIA A).

Both patient groups will have a multimodal assessment at 1 week, 3 months and 12 months after SCI with MRI and neuropsychological tests.

The group of healthy volunteers will only perform one MRI.

DETAILED DESCRIPTION:
Lesions of the spinal cord induce sensory-motor deficits and have various neuropsychological effects. MRI shows a reduction in the volume of the somatosensory and motor cortices, as well as atrophy of the white matter bundles.

Disturbances in brain activity are observed in several critical areas. Patients may experience cognitive impairment and an increased risk of depression and anxiety. Although deep brain stimulation and transcranial magnetic stimulation have shown positive effects, the efficacy of these treatments remains limited, partly due to insufficient understanding of post-SCI brain changes.

The cognitive and behavioral consequences of spinal cord injury are poorly understood and mainly treated by symptomatic therapies, which are often ineffective and may have side effects.

A better understanding of brain networks and their plasticity after spinal cord injury could facilitate the development of targeted therapies, such as cortical or deep basal ganglia stimulation.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 80
* informed consent
* patient with MCT in the previous week
* clinical neurological examination demonstrating a sensory-motor deficit (the severity of which will define the group to which the patient belongs) associated with MCT.

Exclusion criteria:

* Impossibility of following the patient during the study period
* Consent not obtained (adults, non-emancipated minors, persons unable to give consent, research carried out in emergency situations, etc.),
* Not affiliated to a social security scheme,
* Persons under court protection,
* Other life-threatening systemic impairment,
* Prior cognitive impairment,
* Contraindication to MRI (pacemaker, metallic foreign body, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Sensory-motor and cognitive-behavioural impact at supra-spinal level on multimodal Magnetic Resonance Imaging (MRI) | From enrollment to the end of follow up at 12 months
  The difference in task-based functional supraspinal activation pattern evolution (delta beta, GLM) between patient groups (ASIA B,C,D vs. ASIA E) quantified by the students T-score (corrected for multiple comparison) that is associated to the variability of blood flow between the active (participant performs a task in the MRI) and resting (participant is at rest in the MRI) periods. The activity pattern is described by the size (number of voxels) and localization of activated regions.

SECONDARY OUTCOMES:
Cortical volume in mm3 | From enrollment to the end of follow up at 12 months
  Cortical volume in mm3
Difference in evolution of functional motor patterns | From enrollment to the end of follow up at 12 months
  The difference in task-based functional supraspinal activation pattern evolution (delta beta, GLM) between patients and healthy controls quantified by the students T-score (corrected for multiple comparison) that is associated to the variability of blood flow between the active (participant performs a task in the MRI) and resting (participant is at rest in the MRI) periods. The activity pattern is described by the size (number of voxels) and localization of activated regions.
Montreal Cognitive Assessment score | From enrollment to the end of follow up at 12 months
  The correlation, Pearsons r, between functional activity pattern changes (beta, GLM) and cognitive task performance (Montreal Cognitive Assessment score)
Difference in local resting-state connectivity (ALFF) between groups, quantified by the student T-score (corrected for multiple comparisons) | From enrollment to the end of follow up at 12 months
  Difference in local resting-state connectivity (ALFF) between groups, quantified by the student T-score (corrected for multiple comparisons)
Difference in local resting-state connectivity (ReHo) between groups, quantified by the student T-score (corrected for multiple comparisons) | From enrollment to the end of follow up at 12 months
  Difference in local resting-state connectivity (ReHo) between groups, quantified by the student T-score (corrected for multiple comparisons)
Difference in global resting-state connectivity (global efficiency - theory des graphs) between groups, quantified by the student T-score (corrected for multiple comparisons). | From enrollment to the end of follow up at 12 months
  Difference in global resting-state connectivity (global efficiency - theory des graphs) between groups, quantified by the student T-score (corrected for multiple comparisons).
Difference in anatomical connectivity | From inclusion to the last study visit at 12 months
  Difference in anatomical connectivity (using the fractional anisotropy) between groups, quantified by the student T-score (corrected for multiple comparisons).
Measurement of cognitive-behavioral performance by MoCA test | From inclusion to the last study visit at 12 months
  The Monreal Cognitive Assessment tes( MoCA) is a validated cognition test for the early detection of mild cognitive impairment (MCI). It assesses memory, visuospatial abilities, executive functions, attention, language and orientation. The score is comprised between 0 and 30. A score superior or equal to 26 is normal
Measurement of quality of life by SF-36 | From inclusion to the last study visit at 12 months
  The Medical Outcomes Study 36-item Short-Form Health Survey is a widely used, patient self-administered generic measure created to assess health-related quality of life (HRQoL) in the general population. Each item is scored between 0 to 100. A higher score indicates better quality of life.
Beck Depression Inventory (BDI) | From inclusion to the last study visit at 12 months
  The BDI comprises 21 symptom and attitude items (a short version with 13 items exists), describing a specific behavioral manifestation of depression, graded from 0 to 3 by a series of 4 statements reflecting the degree of severity of the symptom. The score is comprised between 0 to 63. A high score means more severe depression
MADRS: Montgomery-Åsberg depression rating scale | From inclusion to the last study visit at 12 months
  The MADRS scale is widely used to measure changes brought about by treatment for depression. It assesses the severity of symptoms in a wide range of areas, including mood, sleep and appetite, physical and psychological fatigue, and suicidal ideation. The score is comprised between 0 to 60. A score of 30 and more is associated to severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France